CLINICAL TRIAL: NCT05947045
Title: Cognitive Training in the Virtual Reality Setting With Children Undergoing Radiotherapy for Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COGVR; NCI-2023-03975 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-06-07; First posted 2023-07-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor
Keywords: Radiotherapy; Brain tumor; Cognitive training; Virtual Reality; Working memory
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPad Cogmed Training (Active Comparator): The investigator will be randomizing participants to complete Cogmed training on an iPad.
  Interventions: Other: Cognitive training via iPad
- Virtual Reality Cogmed Training (Experimental): The investigator will be randomizing participants to complete Cogmed training in Virtual Reality.
  Interventions: Other: Cognitive training via virtual reality

INTERVENTIONS:
Other: Cognitive training via iPad — Participants will complete five sessions of the Cogmed training program on an iPad. Participants will complete sessions over the course of one to two weeks while on campus for radiotherapy. Each session will take place in the Psychology Clinic and consist of 15 to 20 minutes of Cogmed training.
  Arms: IPad Cogmed Training
Other: Cognitive training via virtual reality — Participants will complete five sessions of the Cogmed training program within virtual reality. Participants will complete sessions over the course of one to two weeks while on campus for radiotherapy. Each session will take place in the Psychology Clinic and consist of 15 to 20 minutes of Cogmed training.
  Arms: Virtual Reality Cogmed Training

SUMMARY:
The objective of this study is to estimate the feasibility and acceptability of cognitive training in the virtual reality setting with children undergoing radiotherapy for brain tumors. To achieve this goal, the investigators plan to study children undergoing radiotherapy for brain tumors randomly assigned to cognitive training administered via an iPad or virtual reality. Both groups will also participate in cognitive testing and exams using functional near infrared spectroscopy (fNIRS) pre- and post-intervention. The questions to be investigated are:

1. Will cognitive training via virtual reality be feasible and acceptable for children undergoing radiotherapy for brain tumors as indicated by participation rates, adherence and frequency of side effects?
2. Will cognitive training via virtual reality provide neurocognitive benefits?
3. Will there be predictable changes in brain activity as measured by neuroimaging?

Findings from this study will be used to develop a larger, definitive trial with direct potential to improve cognitive outcomes for children treated for cancer using a safe and effective alternative to desktop- or laptop-based computerized cognitive interventions with great promise for improving quality of life.

DETAILED DESCRIPTION:
The objectives of this study are:

Primary Objective:

• To estimate the participation rate, intervention adherence, and side effects of cognitive training in the virtual reality setting with children undergoing radiotherapy for brain tumors.

Secondary Objectives:

* To estimate the effect size of change in cognitive outcomes associated with cognitive training in the virtual reality setting relative to cognitive training on an iPad.
* To evaluate patterns of cortical activation (oxygenated and deoxygenated hemoglobin responses) pre- and post- cognitive training in the virtual reality setting and on an iPad.

The investigators will use a randomized, single blind (psychology examiner), parallel group design (cognitive training via iPad versus virtual reality) to test hypotheses about behavioral and neurophysiological changes associated with cognitive training in childhood cancer survivors. The investigators will recruit patients who are being treated for a BT with radiotherapy. Patients will participate in study sessions in the Psychology Clinic during routine visits to St. Jude for radiotherapy. fNIRS studies will be conducted with participants randomized to both the virtual reality and iPad groups pre- and post- Cogmed training sessions. The time period between pre- and post-cognitive assessments will be 2 to 4 weeks for both virtual reality and iPad groups.

Participants will be enrolled until 30 patients initiating radiotherapy for a BT are evaluable, with approximately 20 randomized to the virtual reality group and 10 to the iPad group. The investigators expect to recruit and screen up to 45 patients to ascertain 30 eligible participants.

Enrollment and assessment will be completed approximately 18 months after the study begins. Imaging data will be processed approximately two years after the study begins, and study findings will be disseminated within three years after the study begins.

Data management and statistical analysis will be provided locally by the Department of Psychology, the Neuroimaging Division of Radiological Sciences and the Biostatistics Department at St. Jude Children's Research Hospital

ELIGIBILITY:
Inclusion Criteria:

* Initiating radiotherapy for a BT
* Between 8-22 years of age at the time of enrollment
* English or Spanish as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines
* Participant willing to take part in required aspects of Cogmed training

Exclusion Criteria:

* Significant impairment in global intellectual functioning (estimated or full scale IQ < 70 based on standardized testing routinely conducted on primary treatment protocols or as part of the New Oncology Program in Psychology [NOPP])
* History of significant neurological disease preceding BT diagnosis including stroke or head injury with loss of consciousness
* Major sensory or motor impairment that would preclude valid cognitive testing secondary to inability to complete study procedures (e.g., blindness, paresis, poorly controlled seizures/photosensitive epilepsy, inadequate balance to sit or stand unassisted to complete cognitive training)
* Psychiatric condition that would preclude or take precedence over study participation (e.g. active psychosis, suicidal ideation)
* Need for general anesthesia during radiation therapy (note: can participate if only sedated for simulation/planning but not daily treatment)

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Participation Rate | After approach for enrollment, an average of 3 weeks after starting radiation therapy
  The participation rate of this study (i.e., how many patients agree to participate/how many patients are approached for participation) and its 90% Blyth-Still-Casella exact binomial confidence intervals will be estimated for all participants.
Adherence | At the completion of radiation therapy, an average of 6 weeks after enrollment
  The completion of cognitive training sessions is defined as completion of four out of five planned sessions. The rate of completion of cognitive training sessions and its 90% Blyth-Still-Casella exact binomial confidence intervals will be estimated for all participants, and separately for virtual reality and iPad administration groups.
Side Effects | At the completion of radiation therapy, an average of 6 weeks after enrollment
  Summary statistics, including counts and percentages of side effects/cyber sickness symptoms will be provided at pre-, immediate-, and 1-hour post-cognitive training for participants completing training via the iPad or virtual reality.

SECONDARY OUTCOMES:
Neurobehavioral | After completion of post-training assessment, an average of 8 weeks after enrollment
  To estimate the effect size of change in cognitive outcomes associated with cognitive training in the virtual reality setting relative to cognitive training on an iPad. The effect size of the change in cognitive outcomes is defined as the difference in group means/standard deviation (e.g., Cohen's d). The effect size will be calculated separately for change in cognitive outcomes for cognitive training in the virtual reality setting or on iPad. The effect size of the difference of the change between two groups will also be estimated.
Cerebral Hemodynamics | After completion of post-training assessment, an average of 8 weeks after enrollment
  To evaluate patterns of cortical activation (oxygenated hemoglobin response) pre- and post- cognitive training on the iPad and in the virtual reality setting. The effects of VR and iPad based cognitive training will be assessed by n-back and grid-based spatial working memory tasks in conjunction with fNIRS brain imaging of the prefrontal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Heitzer, PhD, ABPP-CN, Principal Investigator — St. Jude Children's Research Hospital; Heather Conklin, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042...